CLINICAL TRIAL: NCT00629707
Title: Cerebral Edema in Pediatric Diabetic Ketoacidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01NS048610 (NIH); R01NS052619-01 (NIH); R01NS052592-01 (NIH)
Record Dates: First submitted 2008-03-04; First posted 2008-03-06 (Estimated); Results first posted 2012-09-12 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Diabetic Ketoacidosis
Keywords: diabetic ketoacidosis; DKA; cerebral edema; brain edema
MeSH Terms: conditions — Diabetic Ketoacidosis; Brain Edema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Slower infusion rate: Patients in this arm will receive an initial intravenous fluid bolus of 10cc/Kg followed by rehydration calculated to replace a deficit of 7.5% of body weight over 48 hours.
  Interventions: Other: intravenous fluid treatment
- 2 (Active Comparator): More rapid infusion: Patients in this arm will receive an initial bolus of 20 cc/Kg of intravenous fluids followed by replacement of an estimated deficit of 10% of body weight over 36 hours plus replacement of 1/2 of urine output volume.
  Interventions: Other: intravenous fluid treatment

INTERVENTIONS:
Other: intravenous fluid treatment — infusion of intravenous fluids (0.9% saline and 0.45% saline)

SUMMARY:
The purpose of this trial is to compare two different rates of fluid administration during diabetic ketoacidosis (DKA) treatment in children to determine which fluid administration rate is more beneficial for brain metabolism and for preventing or decreasing brain swelling during DKA.

DETAILED DESCRIPTION:
Cerebral edema (swelling of the brain) is the most frequent serious complication of diabetic ketoacidosis (DKA) in children. The cause of cerebral edema during DKA is not well understood. Recent studies suggest that it may result from lack of adequate blood flow to the brain during DKA, before treatment starts. Brain injury, resulting in edema, may occur before treatment because of lack of adequate blood flow to the brain and additional injury may occur when adequate blood flow is re-established during treatment (called reperfusion injury). Because additional injury may occur during treatment, it is important to understand whether the rate of administration of intravenous fluids, and, therefore, the speed of reperfusion of the brain, is related to the degree of brain swelling and injury. Most current treatment protocols indicate that intravenous fluids should be administered slowly, but it may be possible that brain injury and swelling might be lessened if adequate blood flow is established more quickly.

In this study, researchers will use magnetic resonance (MR) imaging to compare two different rates of fluid administration during DKA treatment in children. The investigators will use MR imaging to measure brain swelling and metabolism at three time points-twice during treatment and once after recovery from DKA-and will compare these measurements to determine which fluid administration rate has more beneficial effects on brain metabolism and brain swelling.

The study's researchers hypothesize that more rapid re-establishment of blood flow to the brain (via more rapid administration of intravenous fluids) will result in less brain swelling and injury than slower rehydration with delayed re-establishment of adequate brain blood flow will.

ELIGIBILITY:
Inclusion Criteria:

* age 8-18 years
* diagnosis of diabetic ketoacidosis
* able to cooperate with MR scanning

Exclusion Criteria:

* pre-existing cerebral injury or brain structural abnormality
* dental hardware or other metal devices which would interfere with MR imaging

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2008-06; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Glaser, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Medical Center, 2315 Stockton Blvd, Sacramento, California, United States

REFERENCES:
- [Derived] Trainor JL, Glaser NS, Tzimenatos L, Stoner MJ, Brown KM, McManemy JK, Schunk JE, Quayle KS, Nigrovic LE, Rewers A, Myers SR, Bennett JE, Kwok MY, Olsen CS, Casper TC, Ghetti S, Kuppermann N; Pediatric Emergency Care Applied Research Network (PECARN) FLUID Study Group. Clinical and Laboratory Predictors of Dehydration Severity in Children With Diabetic Ketoacidosis. Ann Emerg Med. 2023 Aug;82(2):167-178. doi: 10.1016/j.annemergmed.2023.01.001. Epub 2023 Apr 5. PMID 37024382
- [Derived] Rewers A, Kuppermann N, Stoner MJ, Garro A, Bennett JE, Quayle KS, Schunk JE, Myers SR, McManemy JK, Nigrovic LE, Trainor JL, Tzimenatos L, Kwok MY, Brown KM, Olsen CS, Casper TC, Ghetti S, Glaser NS; Pediatric Emergency Care Applied Research Network (PECARN) FLUID Study Group. Effects of Fluid Rehydration Strategy on Correction of Acidosis and Electrolyte Abnormalities in Children With Diabetic Ketoacidosis. Diabetes Care. 2021 Sep;44(9):2061-2068. doi: 10.2337/dc20-3113. Epub 2021 Jun 29. PMID 34187840
- [Derived] Kuppermann N, Ghetti S, Schunk JE, Stoner MJ, Rewers A, McManemy JK, Myers SR, Nigrovic LE, Garro A, Brown KM, Quayle KS, Trainor JL, Tzimenatos L, Bennett JE, DePiero AD, Kwok MY, Perry CS 3rd, Olsen CS, Casper TC, Dean JM, Glaser NS; PECARN DKA FLUID Study Group. Clinical Trial of Fluid Infusion Rates for Pediatric Diabetic Ketoacidosis. N Engl J Med. 2018 Jun 14;378(24):2275-2287. doi: 10.1056/NEJMoa1716816. PMID 29897851

RESULTS

PARTICIPANT FLOW:
Groups:
- Slow Fluid Infusion: Slower infusion rate: Patients in this arm will receive an initial intravenous fluid bolus of 10cc/Kg followed by rehydration calculated to replace a deficit of 7.5% of body weight over 48 hours.
- Rapid Fluid Infusion: More rapid infusion: Patients in this arm will receive an initial bolus of 20 cc/Kg of intravenous fluids followed by replacement of an estimated deficit of 10% of body weight over 36 hours plus replacement of 1/2 of urine output volume.
Period: Overall Study
Arm/Group | Slow Fluid Infusion | Rapid Fluid Infusion
Started | 10 | 10
Completed | 10 | 8
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Slow Fluid Infusion | Rapid Fluid Infusion | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 10 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 14.2 (3.4) | 11.4 (1.8) | 12.9 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Edema Measured by MR Imaging (Apparent Diffusion Coefficient)
Description: In both groups, brain Apparent Diffusion Coefficient (ADC) measures at 3-6 hours and 9-12 hours after beginning DKA treatment were averaged to determine overall brain ADC during DKA treatment. The brain ADC indicates the distribution of water in the brain and is an indicator of brain swelling (edema). The overall brain ADC values during DKA treatment were compared with the brain ADC measured after recovery to assess the degree of brain edema formation during DKA treatment. The difference in brain ADC, calculated as the averaged treatment values minus the recovery value, was used as the main outcome measure to indicate the degree of brain edema formation
Time Frame: twice during DKA treatment, once at 3-6 hours and at 9-12 after treatment. A normal comparison measurement will be done after recovery from DKA, at least 72 hours after treatment
Population: Data from all enrolled participant that completed the study were analyzed.
Measure: Mean (Standard Deviation); unit: mm^2/sec
Arm/Group | Slow Fluid Infusion | Rapid Fluid Infusion
Number analyzed (Participants) | 10 | 8
mm^2/sec | 36 (30) | 48 (41)

2. Secondary Outcome: Brain NAA/Creatine Ratio & Brain Lactate Measured by MR Spectroscopy, Cerebral Blood Flow & Oxygen Saturation Measured by MR Perfusion Weighted Imaging & Near Infrared Spectroscopy, Mental Status Evaluated by Glasgow Coma Scale Scores.
Time Frame: as for outcome 1
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Slow Fluid Infusion | Rapid Fluid Infusion
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10
Other Adverse Events (participants affected / at risk) | 0/10 | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Slow Fluid Infusion (N=10) | Rapid Fluid Infusion (N=10)
altered mental status (Nervous system disorders) | 0 (0) | 1 (1) — Alteration in mental status during DKA treatment of sufficient severity for suspicion of clinically-apparent cerebral edema
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Slow Fluid Infusion (N=10) | Rapid Fluid Infusion (N=10)
hypoglycemia (Endocrine disorders) | 0 (0) | 1 (2) — blood glucose level below 70 mg/dL during DKA treatment

LIMITATIONS AND CAVEATS:
Study terminated after enrollment of 20 subjects. Review of data from these subjects showed minimal difference between groups and substantial variability suggesting that a larger sample would be very unlikely to show significant differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No